CLINICAL TRIAL: NCT00446225
Title: Phase III, Multicenter, Open-label, Randomized Trial of Tarceva® vs Chemotherapy in Patients With Advanced NSCLC With Mutations in the TK Domain of the EGFR
Brief Title: Phase III Study (Tarceva®) vs Chemotherapy to Treat Advanced Non-Small Cell Lung Cancer in Patients With Mutations in the TK Domain of EGFR
Acronym: EURTAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EURTAC-SLCG // GECP06/01; 2006-003568-73 (EudraCT Number)
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung; cancer; EGFR; Epidermal Growth Factor Receptor; tyrosine kinase; Tarceva®; Erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Erlotinib Hydrochloride; Carboplatin; Gemcitabine; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Erlotinib (Tarceva)150 mg /day
  Patients will receive treatment until disease progression or unacceptable toxicity.
  For all practical effects a treatment cycle will be defined as three weeks of continuous treatment with erlotinib
  Interventions: Drug: Erlotinib
- B (Active Comparator): 4 cycles of Chemotherapy:
  Cisplatin / Gemcitabine; Cisplatin /Docetaxel; Carboplatin / Gemcitabine; Carboplatin / Docetaxel.
  - Cisplatin plus docetaxel: cisplatin 75 mg/m2 i.v. day 1 and docetaxel 75 mg/m2 i.v.
  day 1. Repeat cycles every 3 weeks.
  - Cisplatin plus gemcitabine: Cisplatin 75 mg/m2 i.v. on day 1 and gemcitabine 1250 mg/m2 on days 1 and 8. Repeat cycles every 3 weeks.
  In the case of patients not eligible for treatment with cisplatin, cisplatin can be replaced by carboplatin. The schedules will be the following:
  Docetaxel 75 mg/m2 day 1 and carboplatin AUC = 6 day 1, every 21 days.
  Gemcitabine 1000 mg/m2 days 1 and 8 and carboplatin AUC = 5 day 1, every 21 days.
  Patients in the chemotherapy arm will receive the treatment until disease progression or unacceptable toxicity occurs, or until a maximum of 4 treatment cycles are given.
  Interventions: Drug: Carboplatin; Drug: Gemcitabin; Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Erlotinib — 150 mg/day Patients will receive treatment until disease progression or unacceptable toxicity.
  For all practical effects a treatment cycle will be defined as three weeks of continuous treatment with erlotinib
  Other Names: Tarceva
  Arms: A
Drug: Carboplatin — Gemcitabine 1000 mg/m2 days 1 and 8 and Carboplatin AUC = 5 day 1, every 21 days.
  Docetaxel (75 mg/m2) /carboplatin (AUC=6); Gemcitabine (1000 mg/m2; day 1 and 8) / Carboplatin (AUC=5)
  Patients in the chemotherapy arm will receive the treatment until disease progression or unacceptable toxicity occurs, or until a maximum of 4 treatment cycles are given.
  Other Names: Paraplatin
  Arms: B
Drug: Gemcitabin — Cisplatin (75 mg/m2) / Gemcitabine (1250 mg/m2; day 1 and 8) Patients in the chemotherapy arm will receive the treatment until disease progression or unacceptable toxicity occurs, or until a maximum of 4 treatment cycles are given.
  Other Names: Gemzar
  Arms: B
Drug: Docetaxel — Cisplatin (75 mg/m2) / Docetaxel (75 mg/m2) Patients in the chemotherapy arm will receive the treatment until disease progression or unacceptable toxicity occurs, or until a maximum of 4 treatment cycles are given.
  Other Names: Taxotere
  Arms: B
Drug: Cisplatin — Cisplatin (75 mg/m2) / Docetaxel (75 mg/m2) Patients in the chemotherapy arm will receive the treatment until disease progression or unacceptable toxicity occurs, or until a maximum of 4 treatment cycles are given.
  Other Names: Platinol
  Arms: B

SUMMARY:
A Phase III, multicenter, open-label, randomized trial of Erlotinib (Tarceva®) versus chemotherapy in patients with advanced NSCLC with mutations in the Tyrosine Kinase (TK) domain of the EGFR.

DETAILED DESCRIPTION:
This is a multicenter, phase III, randomized, open-label clinical trial.

146 patients with a diagnosis of advanced (stage IIIB and stage IV), non-squamous-cell, non-small-cell pulmonary carcinoma not treated previously for their disease with chemotherapy who present mutation in the tyrosine kinase domain of the epidermal growth factor receptor, EGFR will be recluted.

The primary objective is to compare the progression-free survival in both treatment arms of the study (conventional chemotherapy vs. erlotinib) in patients with non-squamous-cell, non-small-cell lung cancer (NSCLC) in advanced stage (stages IIIB and stage IV) who have not received previous chemotherapy for their disease and who present mutations in the tyrosine kinase domain of the epidermal growth factor receptor (EGFR).

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Histologically confirmed diagnosis of NSCLC, non epidermoid, stage IV or IIIB with pleural effusion, or N3 tumours not candidate for thoracic radiotherapy, harbouring deletions in the exon 19 or mutation in the exon 21 in the TK of the EGFR.
* Either measurable or evaluable disease.
* Age > 18 years.
* ECOG performance status < 2.
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function
* Patients must be accessible for treatment and follow-up.
* Patients capable of following an adequate therapeutic compliance
* Women of child bearing potential: negative pregnancy test.
* Patients of both genders at a fertile age, including those women having their last menstruation within the two previous years, must follow effective contraceptive measures.
* Ability to swallow.
* Patients with asymptomatic brain metastasis and stable with medical treatment will be eligible for the study. Patients having received radiotherapy for their brain metastasis prior to the systemic treatment for the NSCLC will be also eligible.
* Absence of gastrointestinal tract problems

Exclusion criteria:

* Pregnant or lactating women.
* Women of child bearing potential having a positive pregnancy test in the basal visit or not accomplishing the test.
* Patients of both genders sexually active (at a fertile age) not following contraceptive measures during the study.
* Prior chemotherapy for metastatic disease. Both prior neoadjuvant and adjuvant chemotherapy allowed provided that completed â‰¥ 6 months before entering the study.
* Prior treatment with EGFR targeted therapies.
* Patients may have received radiotherapy, provided that the irradiated lesion is not the only evaluable lesion for response and completed before entering the study.
* Prior experimental pharmacological agent within the 3 weeks prior to the inclusion of the study.
* Any significant ophthalmologic impairment of the eye surface. Use of contact lenses is not recommended.
* Pre-existing motor or sensorial neurotoxicity grade > 2, according to the NCI-CTC criteria.
* Evidence of spinal cord compression.
* Inability to take oral medication and surgical procedures affecting the absorption or implying intravenous or parenteral feeding.
* Any other severe disease or clinical conditions, as, but not only:

  * Unstable cardiopathy despite treatment, myocardial infarction within the 6 months before entering the study
  * History of significant neurological or psychiatric disorders, including dementia and epileptic seizures.
  * Uncontrolled active infection.
  * Uncontrolled peptic ulcer.
  * Unstable diabetes mellitus or any other contraindication for treatment with corticosteroids.
  * AST and/or ALT > 1.5 x UNL associated to alkaline phosphatase > 2.5 x UNL.
  * Any other underlying severe process affecting the ability to take part in the study.
* Absolute contraindication for steroids.
* Dementia or significant mental disorder interfering the understanding and giving the informed consent.
* History of other malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, radically treated prostatic carcinoma with good prognostic (Gleason = 6). History of other curatively treated malignancy and no evidence of disease within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2007-02-15 (Actual); Primary Completion 2012-04-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Rosell i Costa, MD, Study Chair — Spanish Lung Cancer Group; Luis Paz-Ares, MD, Study Chair — Spanish Lung Cancer Group
Locations (76):
- France (19):
  - Centre Hospitalier Universitaire D'Angers, Angers
  - Hôpital Auguste Morvan, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - Centre Hospitalier Intercommunal, Créteil
  - Hôpital A. Mignot, Le Chesnay
  - Centre Hospitalier Du Mans, Le Mans
  - Centre Oscar Lambret, Lille
  - Hôpital du Cluzeau, Limoges
  - Centre Hospitalier Régional, Longjumeau
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier, Périgueux
  - Centre Hospitalier de La Région D'Annecy, Pringy
  - CHU Rennes Hôpital Ponchaillou, Rennes
  - Centre Hosiptalier Genéral de Roanne, Roanne
  - Institut de Cancérologie de La Loire, Saint-Priest-en-Jarez
  - Hôpital Larrey, Toulouse
- Italy (9):
  - CRO di Aviano, Aviano
  - AO Materdomini, Catanzaro
  - AOU Policlinico G. Martino, Messina
  - AO Monaldi, Napoli
  - Casa di Cura "La Maddalena", Palermo
  - Istituti Fisioterapici Ospitalieri, Roma
  - AO S.Camillo Forlanini, Roma
  - Università di Roma "La Sapienza" Az.Policlinico Umb.I°, Roma
  - PO di SS.ma Annunziata, Sassari
- Spain (48):
  - H. Virgen de los Lirios, Alcoy, Alicante
  - H. Torrevieja Salud, Torrevieja, Alicante
  - ICO - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - H. Marqués de Valdecilla, Santander, Cantabria
  - H. Provincial de Castellón, Castellon, Castellón
  - Hospital Insular Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - F.H.Alcorcón, Alcorcón, Madrid
  - H. Fuenlabrada, Fuenlabrada, Madrid
  - H. Son Dureta, Palma de Mallorca, Mallorca
  - H. Ntra. Sra. de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Complejo Hosp. Univ. Juan Canalejo, A Coruña
  - H.G.U. Alicante, Alicante
  - H. Santa Creu i Sant Pau, Barcelona
  - Instituto Universitario Dexeus, Barcelona
  - H.U.Vall D´Hebrón, Barcelona
  - H. Clinic i Provincial, Barcelona
  - H. Althaia, Barcelona
  - H. Duran i Reynals-ICO, Barcelona
  - H. Reina Sofía, Córdoba
  - H. de Donostia, Donostia / San Sebastian
  - ICO Girona -H. Dr. Josep Trueta, Girona
  - H. Virgen de las Nieves, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - H. Arnau de Vilanova, Lleida
  - Hospital San Millan Y San Pedro, Logroño
  - H. de la Princesa, Madrid
  - H. Gregorio Marañón, Madrid
  - H. Ruber Internacional, Madrid
  - H.U. Puerta de Hierro, Madrid
  - Fundación Jimenez Diaz, Madrid
  - Hospial Clinico San Carlos, Madrid
  - H. La Paz, Madrid
  - H. 12 de Octubre, Madrid
  - H. Ramon y Cajal, Madrid
  - H. Carlos Haya, Málaga
  - H.C.Universitario Virgen de la Victoria, Málaga
  - H. Son Llàtzer, Palma de Mallorca
  - Clinica Rotger, Palma de Mallorca
  - H. Virgen del Rocío, Seville
  - H. Nuestra Sra. de Valme, Seville
  - H.C.U.Valencia, Valencia
  - H. General U. de Valencia, Valencia
  - H. Arnau de Vilanova Valencia, Valencia
  - H. Dr. Peset, Valencia
  - H. Miguel Servet, Zaragoza
  - H. Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Derived] Karachaliou N, Mayo-de las Casas C, Queralt C, de Aguirre I, Melloni B, Cardenal F, Garcia-Gomez R, Massuti B, Sanchez JM, Porta R, Ponce-Aix S, Moran T, Carcereny E, Felip E, Bover I, Insa A, Reguart N, Isla D, Vergnenegre A, de Marinis F, Gervais R, Corre R, Paz-Ares L, Morales-Espinosa D, Viteri S, Drozdowskyj A, Jordana-Ariza N, Ramirez-Serrano JL, Molina-Vila MA, Rosell R; Spanish Lung Cancer Group. Association of EGFR L858R Mutation in Circulating Free DNA With Survival in the EURTAC Trial. JAMA Oncol. 2015 May;1(2):149-57. doi: 10.1001/jamaoncol.2014.257. PMID 26181014
- [Derived] Karachaliou N, Gimenez-Capitan A, Drozdowskyj A, Viteri S, Moran T, Carcereny E, Massuti B, Vergnenegre A, de Marinis F, Molina MA, Teixido C, Rosell R. ROR1 as a novel therapeutic target for EGFR-mutant non-small-cell lung cancer patients with the EGFR T790M mutation. Transl Lung Cancer Res. 2014 Jun;3(3):122-30. doi: 10.3978/j.issn.2218-6751.2014.03.02. PMID 25806291
- [Derived] Costa C, Molina MA, Drozdowskyj A, Gimenez-Capitan A, Bertran-Alamillo J, Karachaliou N, Gervais R, Massuti B, Wei J, Moran T, Majem M, Felip E, Carcereny E, Garcia-Campelo R, Viteri S, Taron M, Ono M, Giannikopoulos P, Bivona T, Rosell R. The impact of EGFR T790M mutations and BIM mRNA expression on outcome in patients with EGFR-mutant NSCLC treated with erlotinib or chemotherapy in the randomized phase III EURTAC trial. Clin Cancer Res. 2014 Apr 1;20(7):2001-10. doi: 10.1158/1078-0432.CCR-13-2233. Epub 2014 Feb 3. PMID 24493829
- See also: Spanish Lung Cancer Group website — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Erlotinib Group: Erlotinib (Tarceva)150 mg /day
  Patients will receive treatment until disease progression or unacceptable toxicity.
  For all practical effects a treatment cycle will be defined as three weeks of continuous treatment with erlotinib
  Erlotinib: 150 mg/day Patients will receive treatment until disease progression or unacceptable toxicity.
  For all practical effects a treatment cycle will be defined as three weeks of continuous treatment with erlotinib
- B: Standard Chemotherapy Group: 4 cycles of Chemotherapy:
  Cisplatin / Gemcitabine; Cisplatin /Docetaxel; Carboplatin / Gemcitabine; Carboplatin / Docetaxel.
  3 week cycles of standard intravenous chemotherapy
  * 75 mg/m² cisplatin plus 75 mg/m² docetaxel on day 1 or
  * 75 mg/m² cisplatin on day 1 plus 1250 mg/m² gemcitabine on days 1 and 8
  Patients who were ineligible for cisplatin treatment received intra venous carboplatin chemotherapy instead:
  * 3 week cycles of carboplatin AUC 6 on day 1 with 75 mg/m² docetaxel on day 1 or
  * 3 week cycles carboplatin AUC 5 on day 1 with 1000 mg/m² gemcitabine on days 1 and 8
  Patients in the chemotherapy arm will receive the treatment until disease progression or unacceptable toxicity occurs, or until a maximum of 4 treatment cycles are given.
Period: Overall Study
Arm/Group | A: Erlotinib Group | B: Standard Chemotherapy Group
Started | 87 | 87
Completed | 86 | 87
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Erlotinib Group | B: Standard Chemotherapy Group | Total
Number analyzed (Participants) | 86 | 87 | 173
Age, Continuous [Median (Full Range); unit: years] | 65 [53 to 82] | 65 [46 to 82] | 65 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 68 | 126
  Male | 28 | 19 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 86 | 85 | 171
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Italy | 11 | 8 | 19
  France | 21 | 18 | 39
  Spain | 54 | 61 | 115
Smoking status [Count of Participants; unit: Participants]
  Never smoked | 57 | 63 | 120
  Previous smoker | 22 | 12 | 34
  Current smoker | 7 | 12 | 19
ECOG Performance Status Scale [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  Participants
    ECOG 0 | 27 | 30 | 57
    ECOG 1 | 47 | 45 | 92
    ECOG 2 | 12 | 12 | 24
    ECOG 3 | 0 | 0 | 0
    ECOG 4 | 0 | 0 | 0
Histological diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma | 82 | 78 | 160
  Bronchoalveolar adenocarcinoma | 0 | 2 | 2
  Large-cell carcinoma | 3 | 1 | 4
  Squamous-cell carcinoma | 1 | 0 | 1
  Pleomorphic carcinoma | 0 | 1 | 1
  Adenosquamous carcinoma | 0 | 1 | 1
  Undifferentiated carcinomas | 0 | 4 | 4
Clinical stage [Count of Participants; unit: Participants] — Staging is a classification where cancer is located, if or where it has spread and whether it's affecting other parts of the body.
  There are 5 stages for NSCLC:
  Stage 0:tumor hasn't grown into nearby normal lung tissues Stage I:small tumor that hasn't spread to any lymph nodes Stage II: medium tumor that hasn't spread to the nearby lymph nodes or N1 Stage III: cancer spread to the lymph nodes but haven't spread to other distant parts of the body Stage IV:cancer has spread to more than 1 area in the other lung, the fluid surrounding the lung or the heart, or distant parts of the body
  Participants
    Stage IIIA | 1 | 0 | 1
    Stage IIIB (malignant pleural effusion) | 6 | 5 | 11
    Stage IV | 78 | 82 | 160
    Stage II C | 1 | 0 | 1
Bone metastasis [Count of Participants; unit: Participants] — Bone metastasis in lung cancer occurs when cancer cells spread from the lungs to the bones. This happens when cancer cells break away from the primary lung tumor, travel through the bloodstream or lymphatic system, and establish new tumors in bone tissue.
  Participants
    Yes | 28 | 29 | 57
    No | 58 | 58 | 116
Brain metastasis [Count of Participants; unit: Participants] — Brain metastasis in lung cancer occurs when cancer cells from the lungs spread to the brain. This is a common complication in advanced-stage lung cancer, particularly with non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC). It happens when cancer cells travel through the bloodstream or lymphatic system and invade brain tissue.
  Participants
    Yes | 9 | 11 | 20
    No | 77 | 76 | 153
Type of EGFR mutation [Count of Participants; unit: Participants] — EGFR (epidermal growth factor receptor) mutations in NSCLC types:
  Exon19 Deletions: It leads to the activation of EGFR contributing to cancer cell growth.
  Exon21 L858R Mutation: It involves a substitution of leucine for arginine and leads to receptor activation promoting tumor growth.
  Exon20 Insertion Mutations: Insertion of small amino acid and are often resistant to EGFR inhibitors.
  T790M Mutation: Associated with resistance to TKIs. Exon19-21 Complex Mutations: Across exon 19 & 21.
  Testing for EGFR mutations is crucial for selecting the appropriate therapy in cancer treatment.
  Participants
    Deletion of exon 19 | 57 | 58 | 115
    L858R mutation in exon 21 | 29 | 29 | 58
    Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free-survival
Description: The time from enrollment in the study to tumor progression or death from any cause (whichever occurs first)
Time Frame: From the date of randomization to the date of last follow up, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Erlotinib Group | B: Standard Chemotherapy Group
Number analyzed (Participants) | 86 | 87
months | 9.4 [7.9 to 12.3] | 5.2 [4.4 to 5.8]
Statistical Analysis 1: Comparison: A: Erlotinib Group vs B: Standard Chemotherapy Group; Test type: Superiority; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.27 to 0.64]

2. Secondary Outcome: Objective Response
Description: The objective response rate is defined as the percentage of patients who attain complete response (CR) or partial response (PR); response will be evaluated following RECIST criteria version 1.0.
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on study.
Time Frame: From the date of randomization to the date of last follow up, assessed up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | A: Erlotinib Group | B: Standard Chemotherapy Group
Number analyzed (Participants) | 86 | 87
percentage of participants
  Complete Response (CR) | 2.3 | 0
  Partial Response (PR) | 62.8 | 16.1
  Stable Disease (SD) | 18.6 | 49.4
  Progressive Disease (PD) | 7 | 12.6
  Missing (No Response Assessment) | 9.3 | 21.8

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time, in months, from the inclusion date to the death date. A patient is censored at the last contact date if he/she does not die.Overall survival will be assessed from the date of enrollment in the study until the date of death from any cause. Patients lost to follow-up will be censured on the date of the last follow-up visit.
Time Frame: From the date of randomization to the date of last follow up, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Erlotinib Group | B: Standard Chemotherapy Group
Number analyzed (Participants) | 86 | 87
months | 33.4 [26.7 to 39] | 29.9 [25 to 32.1]
Statistical Analysis 1: Comparison: A: Erlotinib Group vs B: Standard Chemotherapy Group; Test type: Superiority; p = 0.043, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.36 to 0.99]

4. Secondary Outcome: Molecular Markers Related to EGFR and Study Pathology
Description: The study of mutations in serum (serum DNA). This exploratory analysis was performed to determine whether EGFR mutations can reliably be detected in serum thereby reducing the requirement for invasive techniques as well as to enable detection of mutations in patients where no tumor biopsy samples are available.
Time Frame: At baseline
Population: Intention to treat. Serum sample taken at baseline
Measure: Count of Units; unit: Sample of serum
Units Other Than Participants: Sample of serum
Arm/Group | A: Erlotinib Group | B: Standard Chemotherapy Group
Number analyzed (Participants) | 86 | 87
Number analyzed (Sample of serum) | 86 | 87
Sample of serum
  Mutated | 30 | 29
  Wild type | 24 | 23
  Not enough sample | 32 | 35

ADVERSE EVENTS:
Time Frame: 36 months
Description: The severity of AE will be determined using CTCAE version 3.0
Arm/Group | A: Erlotinib Group | B: Standard Chemotherapy Group
All-Cause Mortality (participants affected / at risk) | 55/86 | 54/87
Serious Adverse Events (participants affected / at risk) | 27/86 | 25/87
Other Adverse Events (participants affected / at risk) | 70/86 | 65/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Erlotinib Group (N=86) | B: Standard Chemotherapy Group (N=87)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sigmoiditis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Erlotinib Group (N=86) | B: Standard Chemotherapy Group (N=87)
Fatigue (General disorders) | 48 (48) | 56 (56)
Rash (Skin and subcutaneous tissue disorders) | 66 (66) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 40 (40)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 15 (15)
Aminotransferase rise (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Neuropathy (Nervous system disorders) | 8 (8) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No